CLINICAL TRIAL: NCT04055896
Title: Team Approach to Polypharmacy Evaluation and Reduction in a Long-Term Care Setting: A Feasibility Randomized Controlled Trial
Brief Title: Team Approach to Polypharmacy Evaluation and Reduction in a Long-Term Care Setting
Acronym: TAPER-LTC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 precautions precluded recruitment in long-term care facilities
Sponsor: McMaster University (Other)
Collaborators: Labarge Optimal Aging (Unknown); Canadian Frailty Network (Other)
Responsible Party: Principal Investigator, Derelie Mangin, Professor; Associate Chair and Director, Research David Braley & Nancy Gordon Chair in Family Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2727 (Amendment)
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Long-term Care; Polypharmacy; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: The study will be an adaptive trial design with two phase.
  * Phase 1 will be an internal pilot to allow for refinement.
  * Phase 2 will be a larger randomized controlled trial after Phase 1 refinement
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard of Care as wait list control. Control group will be offered intervention as part of usual clinical care at 6 months.
- TAPER (Experimental): The intervention is medication reduction. This arm is comprised of:
  1. Medication reconciliation
  2. Identification of patient priorities for care
  3. Identification of medications that are potentially appropriate for discontinuation/dose reduction
  4. Linked pharmacist/family physician consultations with patient to discuss medication with intention to reduce
  5. Identification of medications for trial of discontinuation/dose reduction (shared decision making) Pause of medication and clinical monitoring
  Interventions: Other: Medication Reduction

INTERVENTIONS:
Other: Medication Reduction — Systematic approach to reduction in polypharmacy
  Other Names: Medication discontinuation/dose reduction
  Arms: TAPER

SUMMARY:
Medication side effects and interactions between medications are very common in older adults and are related to negative health outcomes. In this study, the investigators will test a new process aimed at reducing unnecessary medication use and drug side effects in seniors using the best medical evidence and patient preferences for treatment. This study will assess how feasible the implementation of this intervention is within a long-term care facility as well as if it is possible. Participants in two long-term care facilities will participate in this study. Measures will include feasibility outcomes regarding the logistics of the intervention as well as patients outcomes (falls, hospitalizations, and medications) collected before and after implementation. This trial will be a randomized control trial with an adaptive trial design.

DETAILED DESCRIPTION:
There are substantial associations between polypharmacy and reduced function from older adults and this is likely to be important in frail older adults both in long term care and in the community. The reversibility of drug-induced mobility impairment is unclear therefore the investigators plan to investigate signals of any impact of reducing polypharmacy on mobility. The investigators chose the long-term care setting given the presence of complete medication administration records and this patient population's high prevalence of polypharmacy and risk of adverse drug events. TaperMD is an electronic tool for systematic medication reduction that incorporates patient priorities, electronic screening for potentially harmful medicines,supporting evidence tools and a monitoring pathway to support medication reduction. This study will examine the feasibility of this tool in a long-term care setting as well as examine. Participants in two long-term care facilities will participate in this study. Measures will include feasibility outcomes regarding the logistics of the intervention as well as patients outcomes (falls, hospitalizations, and medications) collected before and after implementation. The study will be an adaptive trial design with two phases. Phase 1 will be an internal pilot. This will allow the investigators to re-evaluate and modify outcome measures and processes as necessary. Phase 2 of this trial will allow for continuation after adjustments to the process or design has been made in a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* residing in 2 long-term care facilities in Brampton, ON
* on 5 or more long-term medications
* 70 years of age or older
* adequate English language

Exclusion Criteria:

* terminal illness or other circumstance precluding 6 month study period
* recent (within 12 months) comprehensive medication review

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Successful Discontinuation (Difference in mean number of medications; reduction in dose) | 6 months
  Difference in mean number of medications; number of medications reduced in dose

SECONDARY OUTCOMES:
Difference in level of cognition | Baseline, 6 months
  The Mini Mental Status Examination
Difference in level of quality of life | Baseline, 6 months
  EuroQol five dimensions questionnaire (EQ5D-5L) will measure quality of life. Scores range from 0 (low quality of life) to 1 (high quality of life).
Difference in number of falls | Baseline, 6 months
  Total number of falls resulting in medication consultation or treatment recorded in hospital admission and primary care records, and by patient
Difference in level of sleep | Baseline, 6 months
  The sleep question on the 15-Dimensional (15-D) scale will be used. Scores range from 1 (no sleep problems) to 5 (severe sleep problems).
Changes in medication side effects and symptoms (adverse) | 1-week, 3 months, 6 months
  Patient self-report of appearance (new or worsening) of side effects associated with medications
Changes in medication side effects and symptoms (positive) | 1-week, 3 months, 6 months
  Patient self-report of disappearance (improvement or disappearance) of side effects associated with medications
Difference in number of serious adverse events | 1-week, 3 months, 6 months
  Any event that requires in-patient hospitalization or prolongation of existing hospitalization, causes congenital malformation, results in persistent or significant disability or incapacity, is life-threatening or results in death (Health Canada (2011) Guidance Document for Industry - Reporting Adverse Reactions to Marketed Health Products)
Difference in level of physical functioning capacity and ability | Baseline, 6 months
  Time on the timed-up-and-go test
Difference in level of performance of activities of daily living | Baseline, 6 months
  Barthel Index will be used to measure performance of activities of daily living. Ten activities are scored in terms of level of independence or assistance, with higher scores reflecting higher level of independent performance.
Difference in level of frailty | Baseline, 6 months
  The total score on the Edmonton Frail Scale will be used to measure frailty. The scale included 11 items, with scores ranging from 0 (not frail) to 17 (severe frailty).
Difference in level of healthcare utilization use (hospitalizations) | Baseline, 6 months
  Number of hospitalizations
Difference in level of healthcare utilization use (emergency department visits) | Baseline, 6 months
  Number of emergency department visits
Difference in level of healthcare utilization use (physician visits) | Baseline, 6 months
  Number of physician visits
Enrollment rate | 6 months
  Number of participants that enroll in study relative to number of participant invited to participant
Completion rate | 6 months
  Number of participants that complete 6-month collection relative to number of participants enrolled
Time to complete measures | Baseline, 6 months
  Average duration of data collection appointments
Difference in level of mood | Baseline, 6 months
  The total score on the Geriatric Depression Scale (Short Form) will be used to measure mood. The scale includes 15 yes/no items and score range from 0 to 15, with high scores indicating depression.
Difference in level of concern over falling | Baseline, 6 months
  The score on the Falls Efficacy Scale-International (Short Version) will be used to measure falling-related concerns. The scale includes 7 items, with scores ranging from 7 (no concern) to 28 (severe concern of falling)
Difference in level of pain | Baseline, 6 months
  The Brief Pain Inventory (short form) will be used to measure pain severity (mean of 4 items, rated 0-10) and pain interference (mean of 7 items, rated 0-10). Higher scores represent higher pain severity and interference.
Difference in level of incontinence | Baseline, 6 months
  Frequency of incontinence as recorded in patient electronic medical record

OTHER OUTCOMES:
Loved one's perspective of deprescribing | 6 months
  Perspectives from focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Dee Mangin, MBChB, DPH, FRNZC, MD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Holland Christian Homes - Faith Manor, Brampton, Ontario
  - Holland Christian Homes - Grace Manor, Brampton, Ontario